CLINICAL TRIAL: NCT03170284
Title: A Multi-Center Observational Survey of the Efficacy and Safety of Avastin in Addition to Platimun-Based Chemotherapy for First-Line Treatment of Patients With Locally Advanced, Metastatic or Recurrent Non-Small Cell Lung Cancer Other Than Predominantly Squamous Cell Histology
Brief Title: Observational Study to Evalute the Efficacy and Safety of Avastin (Bevacizumab) in Addition to Platinum-Based Chemotherapy for First-Line Treatment of Participants With Non-Small Cell Lung Cancer
Acronym: AVALANCHE
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML21783
Record Dates: First submitted 2017-05-26; First posted 2017-05-31 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bevacizumab: Participants with advanced (stage IIIB/IV) NSCLC other than predominantly squamous cell histology receiving Bevacizumab in accordance with the summary product characteristics (SPC) is observed.
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab is prescribed by physicians as per SPC.
  Other Names: Avastin

SUMMARY:
The purpose of this study is to examine the efficacy of Bevacizumab in addition to platinum-based chemotherapy for first-line treatment of participants with advanced stage (IIIB/IV) non-small cell lung cancer (NSCLC) other than predominantly squamous cell histology.

ELIGIBILITY:
Inclusion Criteria:

In accordance with the SPC. Most important criteria:

* Histology or cytology proven inoperable, locally advanced,metastatic or recurrent (stage IIIB/IV) NSCLC other than predominantly squamous cell histology
* First-line treatment is indicated
* No previous treatment with Bevacizumab

Exclusion Criteria:

In accordance with the SPC. Most important criteria:

* Hypersensitivity to the active ingredient or to any of the excipients
* Hypersensitivity to products derived from Chinese hamster ovary (CHO) cells or to other recombinant human or humanized antibodies
* Pregnancy
* Bevacizumab is contraindicated in the presence of untreated central nervous system metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with locally advanced, metastatic or recurrent non-small cell lung cancer other than predominantly squamous cell histology needing first-line treatment is observed.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2008-06-17 (Actual); Primary Completion 2012-08-01 (Actual); Study Completion 2012-08-01 (Actual)

PRIMARY OUTCOMES:
Time to Disease Progression | up to 45 months
  Time to progression is the time elapsed from the date of enrollment to the first documented progression or to death of any cause. For participants who don't show progression or die until the end of treatment, the date of last contact is taken as the censoring time.

SECONDARY OUTCOMES:
Best Tumor Response | Up to 45 months
  Best tumor response is evaluated as percentage of participants with complete remission (CR), partial response (PR), stable disease (SD) and progressive disease.
Overall Survival | Up to 45 months
  Overall survival is the time elapsed between enrollment and death of any cause. For participants who don't die until the end of treatment, the overall survival data will be analyzed retrospectively based on their date of death after the end of study.
Number of Participants with Serious Adverse Events (SAEs) and Adverse Events (AEs) | Up to 45 months
  An adverse event is any untoward medical occurrence in a patient administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (33):
- Hungary (33):
  - Ogyi, Orszagos Gyogyszereszeti Intezet, Budapest
  - Szent Imre Hospital; Dept. of Oncology, Budapest
  - Orszagos Koranyi TBC es Pulmonologiai Intezet, Budapest
  - Orszagos Onkologial Intezet; Onkologiai Osztaly X, Budapest
  - Semmelweis Egyetem X; Pulmonologiai Klinika, Budapest
  - Uzsoki Utcai Korhaz; Ii. Belgyogyaszat, Budapest
  - Debrecen Uni Medical School; Dept of Pulmonary Medicine, Debrecen
  - Hajdú-Bihar Megyei Önkormányzat Kenézy Gyula Hospital; Infektology Department, Debrecen
  - Csongrad Megyei Onkormanyzat Mellkasi Betegsegek Szakkorhaza, Deszk
  - Koch Robert Korhaz, Edelény
  - Megyei Tudogyogyintezet - Pulmonologia, Farkasgyepű
  - Hospital of Aladar Petz; Dept of Oncoradiology, Győr
  - Petz Aladár County Teaching Hospital; 2nd Department of Psychiatry, Győr
  - Bekes Megyei Tudokorhaz; I. Tudobelosztaly, Gyula
  - Békés Megyei Pándy Kálmán Kórház; Onkologiai tanszek, Gyula
  - Kaposi Mor County Hospital; Dept. of Oncology, Kaposvár
  - Bacs-Kiskun Megyei Korhaz, SZTE AOK Oktato Korhaza, Onkoradiologiai Kozpont, Kecskemét
  - Matrai Állami Gyógyintézet ; Bronchológia, Mátraháza
  - Szent Ferenc Kórház; Belgyógyászat, Miskolc
  - Karolina Korhaz, Mosonmagyaróvár
  - Josa Andras Korhaz; Dept of Oncoradiology, Nyíregyháza
  - Szabolcs-Szatmar-Bereg County Josa Andras Hospital; 1St Depatment of Pulmonary Medicine, Nyíregyháza
  - Pécsi Tudományegyetem Áok; Onkoterapias Intezet, Pécs
  - Baranya County Hospital; Pulmonology Dept, Pécs
  - Sopron Megyei Jogu Varos Erzsebet Korhaza Mellkasgyogyaszat, Sopron
  - Tolna Megyei Balassa Janos Korhaz; Iv. Belgyogyaszati Osztaly, Szekszárd
  - Fejér Megyei Szent György Kórház; Pulmonary Medicine, Székesfehérvár
  - Jász-Nagykun-Szolnok Megyei Hetényi Géza Kórház; Onkológiai Osztály, Szolnok
  - Vas Megyei Markusovszky Korhaz ; Oncoradiology, Szombathely
  - Vas Megyei Markusovszky Korhaz ; Pulmonology, Szombathely
  - Komarom-Esztergom Megyei Onkormanyzat Szent Borbala Korhaz; Haematologiai Osztaly, Tatabánya
  - Inst. of Pulmonary Medicine, Torokbalint; 2Nd Dept of Pulmonary Medicine, Törökbálint
  - Zala Megyei Korhaz; Dept of Pulmonary Medicine, Zalaegerszeg

REFERENCES:
- [Derived] Tolnay E, Ghimessy AK, Juhasz E, Sztancsik Z, Losonczy G, Dombi P, Vennes Z, Helf L, Csada E, Sarosi V. The efficacy and safety of bevacizumab in addition to platinum-based chemotherapy for the first-line treatment of patients with advanced nonsquamous non-small-cell lung cancer: Final results of AVALANCHE, an observational cohort study. Oncol Lett. 2019 Feb;17(2):1750-1760. doi: 10.3892/ol.2018.9766. Epub 2018 Nov 27. PMID 30675234